CLINICAL TRIAL: NCT06889545
Title: Evaluation of a Feasible Frailty Assessment Tool for Preoperative Risk Evaluation of Older Patients
Brief Title: Comparison of Preoperative Frailty Assessment Tools
Acronym: PREFAS
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-101410-BO-ff
Record Dates: First submitted 2025-02-23; First posted 2025-03-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Frailty in Older Adults; Frailty/Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older patients: Patients at 70 years and above scheduled for surgery
  Interventions: Other: Assessment of frailty using multiple tools

INTERVENTIONS:
Other: Assessment of frailty using multiple tools — This is an observational study without any intervention. Frailty is assessed using multiple tools and postoperative outcome is compared.

SUMMARY:
Frailty is a significant risk factor for postoperative complications and functional decline. Preoperative assessment of frailty is therefore recommended in all older adults. However, despite the availability of many frailty tools, few have been tested in the preoperative setting and there is little comparison of their predictive value in identifying patients at risk. The aim of this study is to investigate which of the following instruments for determining frailty has the highest predictive power with regard to the occurrence of postoperative complications: Risk Analysis Index, Clinical Frailty Scale, the Groningen Frailty Indicator, the Edmonton Frail Scale and the LUCAS-FI. The aim of this research project is to identify a suitable frailty instrument for preoperative risk stratification of older patients during the premedication visit.

ELIGIBILITY:
Inclusion Criteria:

* 70 years and older
* scheduled surgery
* estimated time of surgery 120 Minutes or more

Exclusion Criteria:

* insufficient German language skills (for cognitive testing)
* mental retardation
* relevant psychiatric disorder (not allowing for cognitive testing)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of the Medical University Centre Hamburg, Germany
Sampling Method: Non-Probability Sample
Enrollment: 584 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Complications in the first 30 days after surgery | 30 days
  Measured by Clavien-Dindo classification

SECONDARY OUTCOMES:
Functional state (activities of daily living) | one, three and six months after surgery
  Measured using WHO Disability Assessment Schedule 2.0
Postoperative Quality of Recovery | postoperative day 2
  Measured by Quality-of-Recovery-15 questionnaire
Muscle loss during hospitalisation | From date of enrollment, up to 4 weeks after surgery
  measured by bioimpedance prior to admission and before discharge from hospital
Postoperative delirium | postoperative day 1 to 5
  Measured by 3D-Confusion Assessment Method
Length of stay | from day of surgery, up to 4 weeks after surgery
  days spent in hospital after surgery
Discharge destination | up to 4 weeks after surgery
  e.g.:home, nursing home, other hospital
Cognitive state | 3 and 6 months after surgery
  Using 5-Minute Montreal Cognitive Assessment (telephone-MOCA). A maximum of 15 points and a minumum of 0 points can be archieved; a higher score indicates better cognitive performance.
Quality-of-Life (QoL) | 3 and 6 months after surgery
  Measured by WHO-Quality of Life in older adults (WHOQOL-OLD) questionnaire. The WHOQOL-OLD is evaluated by calculating scores for its six facets and summing them, with higher scores indicating a better perceived quality of life.
Frailty progression measured by LUCAS-FI | 3 and 6 months after surgery
  Frailty assessment with Longitudinal Urban Cohort Aging Study Functional Index (LUCAS-FI)-questionnaire (telephone interview) The LUCAS-FI is evaluated by integrating both risk factors and protective resources, with the balance between them determining the degree of frailty.
Frailty progression measured by GFI (questionnaire) | 3 and 6 months after surgery
  frailty assessment with Groningen Frailty Indicator (GFI) questionnaire (telephone interview).
  The GFI is evaluated by summing its item responses, with higher scores indicating a higher degree of frailty.
Frailty progression measured by EFS | 3 and 6 months after surgery
  Frailty assessment by Edmonton Frail Scale (EFS), (score filled by physician, patient telephone interview).
  1 to 10 points can be archieved, more points indicate a greater level of frailty.
Frailty progression by RAI measurement. The Risk Analysis Index (RAI) is evaluated by summing weighted risk factors and protective variables, with higher scores indicating greater patient vulnerability. | 3 and 6 months after surgery
  Frailty assessment with Risk Analysis Index (index filled by physician, patient telephone interview)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Cynthia Olotu, MD, Principal Investigator — University Medical Centre Hamburg
Locations (1):
- University Medical Centre Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Strict data protection guidelines prevent patient data from being made available to third parties. In specific cases, anonymised data may be provided after individual examination and consultation with the responsible ethics committee.